CLINICAL TRIAL: NCT07226817
Title: A Phase 1, Open-label, Single-site, Multi-part, Non-randomized, Parallel-group Study to Assess the Relative Bioavailability of BMS-986435 Tablet Formulations (Parts 1 & 2) and Food Effect on the Selected BMS-986435 Tablet Formulation (Part 3) in Healthy Adult Participants
Brief Title: A Study to Assess the Relative Bioavailability of BMS-986435 and Food Effect on the BMS-986435 in Healthy Adult Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV029-1024
Record Dates: First submitted 2025-11-07; First posted 2025-11-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Treatment A (Experimental)
  Interventions: Drug: BMS-986435
- Treatment B (Experimental)
  Interventions: Drug: BMS-986435
- Treatment C (Experimental)
  Interventions: Drug: BMS-986435
- Treatment D (Experimental)
  Interventions: Drug: BMS-986435
- Treatment E (Experimental)
  Interventions: Drug: BMS-986435
- Treatment F (Experimental)
  Interventions: Drug: BMS-986435
- Treatment G (Experimental)
  Interventions: Drug: BMS-986435

INTERVENTIONS:
Drug: BMS-986435 — Specified dose on specified days
  Other Names: MYK-224

SUMMARY:
This study is designed to evaluate the relative bioavailability (rBA) of multiple test tablet formulations of BMS-986435 compared to an equal dose of the BMS-986435 reference tablet formulation. The effect of food on the selected BMS-986435 tablet formulation will also be evaluated.

ELIGIBILITY:
Inclusion Criteria

* Participants must have a body weight of ≥ 45 kg and BMI between 18 and 32 kg/m2, inclusive
* Participants must be healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), clinical laboratory assessments
* Participants must have documented left ventricular ejection fraction (LVEF) ≥ 60% and absence of significant cardiac abnormality at screening, as determined by local transthoracic echocardiogram (TTE) assessment
* Other protocol-defined Inclusion/Exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to Day 28
Area under the concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to Day 28
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to Day 28

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve truncated at 72-hour (AUC(0-72h)) | Up to Day 28
Time of maximum observed concentration (Tmax) | Up to Day 28
Half-life (T-HALF) | Up to Day 28
Apparent total body clearance (CLT/F) | Up to Day 28
Volume of distribution of terminal phase (Vz/F) | Up to Day 28
Number of participants with Adverse Events (AEs) | Up to Day 35
Number of participants with Serious AEs (SAEs) | Up to Day 35
Number of participants with clinical laboratory abnormalities | Up to Day 28
Number of participants with vital sign abnormalities | Up to Day 28
Number of participants with physical examination abnormalities | Up to Day 28
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07226817.html